CLINICAL TRIAL: NCT07134439
Title: Identifying Fundamental Mechanisms of Skeletal Muscle Ageing in Older Men Undergoing Androgen Deprivation Therapy: a Feasibility Study
Acronym: MASS-ADT
Status: Not yet recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 353219
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Sarcopenia; Prostate Cancer; Muscle Atrophy; Androgen Deprivation Therapy
MeSH Terms: conditions — Sarcopenia; Prostatic Neoplasms; Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, muscle biopsy samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men undergoing Androgen Deprivation Therapy for the treatment of prostate cancer

SUMMARY:
To find out whether it is possible to run a study looking at the underlying markers of ageing in muscle quality and quantity in men receiving Androgen Deprivation Therapy for prostate cancer treatment.

To determine the feasibility of conducting an observational study examining the association of fundamental biological markers of ageing with changes in body composition and skeletal muscle morphology following ADT in older men undergoing prostate cancer treatment.

DETAILED DESCRIPTION:
Androgen Deprivation Therapy (ADT) is a well-established therapy for prostate cancer that improves overall survival rates, reduced rates of metastatic prostate cancer and death from prostate cancer . ADT is most commonly delivered through medical castration. It works due to the sensitivity of prostate cancer to androgen signalling. Gonadotropin-releasing hormone (GnRH) agonists or antagonists are used to lower systemic testosterone and oestrogen levels and thereby control the prostate cancer. However, the reduction of these hormones can lead to systemic side-effects including changes in body composition such as increased fat mass and reduced muscle mass and subsequently result in sarcopenia and metabolic side-effects.

Sarcopenia is a condition underpinned by profound reductions in muscle mass and quality that occur in such sufficient magnitude as to lead to impairments in muscle function, independence and mobility. Moreover, sarcopenia is known to increase risk of falls, lead to impairments in quality of life, and increase mortality (independent of activities of daily living, age, and other factors). Resistance exercise is the gold standard treatment for sarcopenia, although this non-pharmacological stimulus has been shown to increase testosterone levels. Despite the potential rise in testosterone levels, resistance exercise has been shown to improve prostate cancer-specific mortality as well as providing functional benefits. Thus, additional downstream pathways are likely upregulated during the ageing process in older men undergoing Androgen Deprivation Therapy .

Ageing is a heterogenous process characterised by cellular senescence, telomere shortening, systemic inflammation and mitochondrial dysfunction and other "hallmarks of ageing". In animal models it has been shown that targeting these processes can extend healthspan and reduce the development of age-related conditions. There are small scale studies in humans trialling the use of drugs that target these ageing processes, known as geroprotectors. However, the fundamental mechanisms underpinning skeletal muscle atrophy and changes in body composition in patients undergoing ADT for prostate cancer are not well understood.

This study will assess the feasibility and acceptability of an observational cohort study to identify the fundamental mechanisms by which ADT is associated with changes in body composition following ADT in older adults with prostate cancer. Older adults are the focus of this study as the risk of side effects from ADT increases with age and the older population is poorly represented in research, including in research with prostate cancer populations . By identifying what processes may be involved in muscle atrophy following ADT, we will be able to better understand how to prevent this occurring and potentially target these pathways using geroprotectors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years old at time of recruitment
* Able to provide informed consent to participate
* Known prostate cancer due to be initiated on ADT for the first time (with or without Androgen Receptor Targeted Agents (ARTA) or radiotherapy), or initiated within two weeks prior to recruitment.
* Individuals involved in other research will be eligible to participate so long as the other research does not involve potential changes to the standard ADT care the participant will be receiving and does not involve an intervention aimed at reducing the muscle atrophy associated with ADT.

Exclusion Criteria:

* Systemic anti-cancer therapy within one year of recruitment (for prostate cancer or any other concomitant cancer)
* Planned surgery (not including eye surgery or other minor surgery) within six months of ADT
* Any other condition previous or current which, in the judgement of the responsible clinician, is likely to interfere with the trial / assessments.
* Lacks capacity to consent

Exclusion criteria for those consenting to optional muscle biopsy:

* On treatment with clopidogrel, high-dose aspirin, dipyridamole or anticoagulants
* Known bleeding disorder or platelets <75x103/mL

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Men >= 65 years old who are starting Androgen Deprivation Therapy for treatment of prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment and retention rate | 6 months

SECONDARY OUTCOMES:
Rectus femoris ultrasound echogenicity at four-six months, adjusting for baseline echogenicity readings. | 6 months
Ultrasound Bilateral Anterior Thigh Thickness (BATT) at four-six months, adjusting for baseline BATT | 6 months
Bilateral anterior thigh subcutaneous tissue thickness at four-six months, adjusting for baseline thickness | 6 months
Skeletal muscle mass (SMM) assessed using bioelectrical impedance analysis (BIA) at four-six months, adjusting for baseline SMM | 6 months
Fat mass from BIA at four-six months, adjusting for baseline fat mass | 6 months
Handgrip strength at four-six months, adjusting for baseline strength | 6 months
Quadriceps strength outcomes using isokinetic dynamometry, adjusting for baseline strength | 6 months
Short physical performance battery (SPPB) at four-six months, adjusting for baseline SPPB | 6 months
Lower limb muscular power measured by the vertical jump test at four-six months, adjusting for baseline power | 6 months
European Organisation For Research And Treatment Of Cancer (EORTC) Core Quality of Life questionnaire score at four-six, adjusting for baseline score. | 6 months
Biological markers of accelerated ageing | 6 months
Frailty level | 6 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riachy R, McKinney K, Tuvdendorj DR. Various Factors May Modulate the Effect of Exercise on Testosterone Levels in Men. J Funct Morphol Kinesiol. 2020 Nov 7;5(4):81. doi: 10.3390/jfmk5040081. PMID 33467296
- [Background] Lopez-Otin C, Blasco MA, Partridge L, Serrano M, Kroemer G. Hallmarks of aging: An expanding universe. Cell. 2023 Jan 19;186(2):243-278. doi: 10.1016/j.cell.2022.11.001. Epub 2023 Jan 3. PMID 36599349
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Cao L, Morley JE. Sarcopenia Is Recognized as an Independent Condition by an International Classification of Disease, Tenth Revision, Clinical Modification (ICD-10-CM) Code. J Am Med Dir Assoc. 2016 Aug 1;17(8):675-7. doi: 10.1016/j.jamda.2016.06.001. No abstract available. PMID 27470918
- [Background] Haseen F, Murray LJ, Cardwell CR, O'Sullivan JM, Cantwell MM. The effect of androgen deprivation therapy on body composition in men with prostate cancer: systematic review and meta-analysis. J Cancer Surviv. 2010 Jun;4(2):128-39. doi: 10.1007/s11764-009-0114-1. Epub 2010 Jan 21. PMID 20091248